CLINICAL TRIAL: NCT05403775
Title: Application of 3D Printing Guide Plate in Transforaminal Epidural Steroid Injection (TFESI) Combined With Pulsed Radiofrequency (PRF) Treatment
Brief Title: Application of 3D Printing Guide Plate in Dorsal Root Ganglion Intervention Treatments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M2022206
Record Dates: First submitted 2022-05-30; First posted 2022-06-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-05

CONDITIONS: Lumbar Disc Herniation; Lumbar Spinal Stenosis
Keywords: Transforaminal epidural steroid injection; Dorsal root ganglion pulsed radiofrequency; 3D printing guide plate; Lumbosacral radicular pain
MeSH Terms: conditions — Intervertebral Disc Displacement; Spinal Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D printing guide plate group (Experimental): 3D-printed customized guide plate will be used to guide the puncture in TFESI combined with dorsal root ganglion PRF.
  Interventions: Other: 3D printing guide plate
- Conventional guidance group (Active Comparator): The surgeons would place the needle according to his/her previous experience under the guidance of C-arm fluoroscopy.
  Interventions: Other: Conventional guidance

INTERVENTIONS:
Other: 3D printing guide plate — 3D-printed customized guide plate will be used to guide the puncture in TFESI combined with dorsal root ganglion PRF to help to reduce intra-operative radiation.
  Arms: 3D printing guide plate group
Other: Conventional guidance — The surgeons would place the needle according to his/her previous experience under the guidance of C-arm fluoroscopy.
  Arms: Conventional guidance group

SUMMARY:
This study applies 3D-printed customized guide plate in assisting the accurate puncture in transforaminal epidural steroid injection (TFESI) combined with pulsed radiofrequency (PRF) treatment. This technique can shorten reduce the intra-operative radiation, and do not affect the surgical outcome.

DETAILED DESCRIPTION:
Lumbar disc herniation (LDH) is a common degenerative spine disease and it can cause low back pain and lumbosacral radicular pain (LSRP). Transforaminal epidural steroid injection (TFESI) is one of the most common minimally invasive interventions for the treatment of LDH. TFESI combined with dorsal root ganglion pulsed radiofrequency (PRF) is an effective procedure for treating LSRP. Needle Puncture is the key technology in this procedure.

In the past when there were no customized guides, the surgeons would place the needle according to his/her previous experience under the guidance of C-arm fluoroscopy or CT. If the position of the needles is not satisfactory, repeated procedure will be performed. This would lead to an increase in the duration of surgery and intra-operative radiation, which is detrimental to both the surgeon and the patient. This problem is well solved by applying the 3D printing guide plate.

The application procedure for the the 3D printing guide plate: the model of the spine is established according to the patient's CT scan data to prepare the customized guide plate, then sterilize them for future use. The final position of needle is confirmed by C-arm fluoroscopy or CT.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old,
2. Chronic lumbosacral radicular pain lasting ≥12 weeks,
3. Dominant leg pain with less intense back pain,
4. The previous failure of conservative management such as physiotherapy, exercise therapy, or analgesic medications,
5. Pain intensity≥4 out of 10 on the numerical rating scale (NRS),
6. Segmental pain of a radicular nature originating from the lumbar segments and with a shooting or lancinating quality corresponding to a dermatome suggestive of the involved nerve root,
7. Availability of computed tomography/magnetic resonance imaging findings of pathology concordant with the side and level of their clinical features.

Exclusion Criteria:

1. Patient refusal to participate in the study,
2. Pregnant or nursing
3. Progressive motor weakness in the affected leg,
4. Allergies to local anesthetics, contrast dyes or steroids
5. Significant anatomic deformity (either congenital or acquired) making it difficult to access the foramen as evidenced by computed tomography/magnetic resonance imaging
6. Presence of cancer accounting for back pain
7. Patients with platelet dysfunction, bleeding disorder or continuing anticoagulant treatment
8. Steroid injection within the previous 12 weeks,
9. Systemic infection,
10. Injection site infection,
11. Unstable medical or psychiatric condition

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07-08 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
C-arm fluoroscopy times | Intraoperative
  Numbers of using C-arm fluoroscopy

SECONDARY OUTCOMES:
Puncture time | Intraoperative
  Time from the first puncture to the last puncture
Numerical rating scale (NRS) | Postoperative 1 day, 1 month, 3 months
  NRS at One day, 1 month, 3 months after the operation
MacNab | Postoperative 3 months
  Patient satisfaction using the modified MacNab criteria
Complications | Intraoperative
  Complication like nerve injury, blood, hemotoma, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Pain medicine center of Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No